CLINICAL TRIAL: NCT01918540
Title: Comparing Hollow and Solid Centralizer Designs When Using a Polished, Collarless, Tapered Hip Prosthesis Stem (MS30). A Prospective, Randomized, Multicenter Study Evaluated by RadioStereometric Analysis (RSA).
Brief Title: Importance of Hollow or Solid Centralizer for Polished, Collarless and Tapered Stems in Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Centralizer study
Record Dates: First submitted 2013-07-04; First posted 2013-08-07 (Estimated); Last update posted 2014-11-26 (Estimated); Status verified 2014-11

CONDITIONS: Total Hip Arthroplasty
Keywords: Radiostereometry; Total Hip Arthroplasty; Stem design

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hollow Centralizer (Active Comparator): The stem used (MS30)was originally designed with a solid centralizer but has been redesigned to be used with a hollow centralizer.
  Interventions: Procedure: Hollow Centralizer; Device: MS-30 femoral stem
- Solid Centralizer (Active Comparator): The stem used (MS30)was originally designed with a solid centralizer but has been redesigned to be used with a hollow centralizer.
  Interventions: Procedure: Solid Centralizer; Device: MS-30 femoral stem

INTERVENTIONS:
Procedure: Hollow Centralizer — The stem used (MS30)was originally designed with a solid centralizer but has been redesigned to be used with a hollow centralizer. The patients are randomized to either solid or hollow centralizer
  Arms: Hollow Centralizer
Procedure: Solid Centralizer — The stem used (MS30)was originally designed with a solid centralizer but has been redesigned to be used with a hollow centralizer. The patients are randomized to either solid or hollow centralizer
  Arms: Solid Centralizer
Device: MS-30 femoral stem — This is the stem used in the study.

SUMMARY:
The study aims at comparing the effect of hollow or solid centralizer designs on the long time fixation behaviour of hip prosthesis stems that are polished, tapered and collarless. In a prospective, controlled and randomized study comprising two groups of 30 patients/hips each, the patients will be followed up by RadioStereometric Analysis (RSA) for ten years. In completion general health questionnaires as well as hip specific scoring instruments will be used to evaluate patient satisfaction and outcome.The hypothesis of the study is that the different centralizers will result in different migration patterns of the stems, which might affect the risk for late aseptic loosening.

ELIGIBILITY:
Inclusion Criteria:

* Primary osteoarthritis of the hip necessitating primary hip replacement
* Charnley classification group A and B
* Age 60 - 85 years old at the inclusion time of the study.

Exclusion Criteria:

* Secondary osteoarthritis
* Rheumatoid arthritis
* Malignant disease
* Severe osteoporosis
* Earlier fracture or operation in the hip to be operated on
* Peroperative fracture
* Ongoing corticosteroid (oral) or immunosuppressive medication
* Personal disorders (dementia, alcohol or drug abuse etc) suspected of making completion of the trial uncertain.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-02; Primary Completion 2004-02 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Radiostereometric Analysis (RSA) | The first postoperative day, 6 months, 1, 2, 5 and 10 years
  This will measure the change in stem migration over time and be indicative of long term result.

SECONDARY OUTCOMES:
x-ray | The first postoperative day, 6 months, 1, 2, 5 and 10 years
  On standard x-rays the progress of radiolucent lines or other signs of loosening will be measured
Hip specific questionnaire | Preoperatively, 1, 2, 5 and 10 years
  Hip disability and Osteoarthritis Score (HOOS) - this is a hip specific questionnaire that will measure how the operation has affected the patients hip function and pain situation
General health questionnaire | Preoperatively, 1, 2, 5 and 10 years
  EuroQol (EQ-5D) - a standardized instrument for use as measure of general health outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopedics, Skane University Hospital, Lund University, Lund, Skåne County, Sweden